CLINICAL TRIAL: NCT06153576
Title: The Value of Systematic Biopsies During Vertebroplasty for the Treatment of Osteoporotic Vertebral Fractures
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Imagerie03
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Vertebral Compression Fracture; Myeloma; Bone Metastases; Malignant Bone Tumour; Lymphoma; Plasmocytoma
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma; Plasmacytoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background : Vertebral fracture is the most common complication of osteoporosis. Vertebroplasty is a widespread treatment modality for osteoporotic vertebral fractures, providing consolidation, rapid pain relief and preventing secondary vertebral collapse. Performing a biopsy at the same time as the operation does not lengthen the procedure or increase the risk of complications. The question therefore arises as to whether it is cost-effective diagnostically: are non-osteoporotic vertebral lesions detected when biopsies are taken? Methods: The investigators carried out a single-centre retrospective study at Nice University Hospital.

From January 2016 to March 2022, 1729 biopsies were performed during 1439 vertebroplasty procedures on 1120 patients.

The pre-operative laboratory work-up included a blood count, a C-reactive protein assay and a coagulation test.

The imaging work-up systematically included MRI, unless contraindicated, in which case CT alone was performed.

Vertebroplasty was performed in an interventional CT suite under dual CT and fluoroscopic guidance. The systematic biopsy sample was then sent to the anatomopathology department for analysis.

Findings :

The samples detected cancer in 35 patients, including 5 (0.44%) for whom the pre-operative work-up had not raised any suspicion.

All the incidental findings were haemopathies, including 4 myelomas and one lymphoma.

Conclusion :

These results highlight the good performance of MRI in distinguishing osteoporotic vertebral fractures from solid tumour metastases.

However, an exhaustive pre-operative work-up does not seem to be able to formally rule out an underlying malignant lesion.

The investigators therefore recommend that biopsies be taken systematically when performing vertebroplasty.

ELIGIBILITY:
Inclusion Criteria:

* all patients who underwent a vertebroplasty with bone biopsy

Exclusion Criteria:

* non-vertebral bone biopsies
* not performed during vertebroplasty

Ages: 17 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent a vertebroplasty with bone biopsy during the study period in the osteoarticular interventional radiology department of the Pasteur 2 hospital of the CHU of Nice
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of incidental discovery of malignant lesions during systematic biopsies for the treatment of vertebral compression fractures | 5 years and 2 months
  incidental findings of neoplasia during vertebroplasty for presumed osteoporotic fractures

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France